CLINICAL TRIAL: NCT00226577
Title: Phase II Study of Neoadjuvant Chemotherapy With Gemcitabine and Pemetrexed in Resectable Non-Small-Cell Lung Cancer (NSCLC) With Pharmacogenomic Correlates.
Brief Title: Pharmacogenomic & Phase II Study of Gemcitabine and Pemetrexed in Non-Small-Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13726; H3E-US-X009 (Other: Eli Lilly & Company)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-01

CONDITIONS: Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; resectable; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Pemetrexed; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre-Surgery Chemotherapy (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Pemetrexed; Procedure: Surgery

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine (GemzarR) 1500 mg/m2
  Other Names: Gemzar®
Drug: Pemetrexed — Pemetrexed (AlimtaR) 500 mg/m2
  Other Names: Alimta®
Procedure: Surgery — When the chemotherapy treatment is completed, the patient's tumor response will be evaluated by a CT scan, pulmonary function test, and another PET scan between days 50 and 63 (during weeks 8 and 9). If there is no growth or spread of the cancer on any of these tests, patients will then proceed to have surgery by week 10 to remove the cancer.

SUMMARY:
This study will evaluate the efficacy and safety of chemotherapy given prior to having lung cancer surgically removed. Patients with resectable non-small cell lung cancer will receive gemcitabine and pemetrexed together for 4 times biweekly. Patients will be seen by a medical oncologist prior to each cycle of chemotherapy given. The medical oncologist will review patient's bloodwork and symptoms prior to approving next cycle of chemotherapy. All patients will then be evaluated with scans to determine response to chemotherapy and to determine if patient is a surgical candidate. These patients will then proceed to surgery to have the lung cancer removed. Follow up visits include bloodwork, scans, and a visit with the medical oncologist every three months for two years, then every six months for three years to monitor for disease recurrence.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of neoadjuvant chemotherapy with gemcitabine and pemetrexed given together 4-times biweekly in patients with resectable NSCLC. All patients will be seen by members of the Thoracic Oncology Program at the H. Lee Moffitt Cancer Center and Research Institute in Tampa, Florida, and they will be discussed in our weekly multidisciplinary thoracic oncology conference. The conference includes pathologists, radiologists, thoracic surgeons, pulmonologists, radiation oncologists, medical oncologists, oncology nurse specialists, case managers, social workers, and clinical trials coordinators. They will have initial tests as outlined in the study timetable. Patients will receive gemcitabine biweekly on days 1, 15, 29, and 43 at a dose of 1,500 mg/m2. They will also receive pemetrexed at a dose of 500 mg/m2 on days 1, 15, 29, and 43. Gemcitabine will be given first over a period of 30 minutes i.v. followed by pemetrexed over 10 minutes i.v. All patients will get a post induction chemotherapy PET scan, CT scan, and PFT's including a DLCO. They will then go on to thoracotomy including bronchoscopy and mediastinal lymph node dissection between days 64 and 77 if the tumor is deemed completely resectable on restaging studies.

The administration of chemotherapy at the earliest time (neoadjuvant or induction chemotherapy) following diagnosis in an effort to reduce the risk of disease recurrence. This approach also allows for investigations of molecular parameters that may affect response to chemotherapy and patients' survival. It is our hypothesis that the expression of genes associated with activation, inactivation, and efficacy of the drugs gemcitabine and pemetrexed will predict response to therapy and prognosis. We further hypothesize that the expression of these genes will be altered during chemotherapy, and that the global assessment of tumor proliferation, apoptosis, and genome damage is associated with response to therapy. We propose a phase II study of neoadjuvant chemotherapy with gemcitabine and pemetrexed in patients with resectable NSCLC, specifically correlating molecular and genetic parameters to the primary clinical study endpoint disease response (radiographic CR+PR) and the secondary endpoints complete pathological response at surgery, disease-free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Microscopically confirmed non-small cell carcinoma of the lung, which may be confirmed at the initial bronchoscopy and mediastinoscopy, or by transthoracic needle biopsy.
* No prior therapy for lung cancer.
* Patients must have disease stages IB (T2N0M0), IIA (T1N1M0), IIB (T2N1M0 and T3N0M0), or IIIA (T3N1M0 and T1-3N2M0). Patients with 2 lesions in one lobe (T4) (Stage IIIB) are eligible.
* Patients must be deemed medically fit for surgical resection by a thoracic surgeon.
* Patients must have an ECOG performance status of Zero or One.
* Patients must have measurable or evaluable disease.
* Measurable Disease: Any mass reproducibly measurable in one diameter (RECIST criteria).
* Evaluable disease: Lesions apparent on chest CT, which do not meet the criteria for measurability. These include ill-defined masses associated with post obstructive changes.
* Age >18 years.
* Patient must be able to understand and sign the informed consent.
* Patients must be >12 weeks from prior major surgery, such as a coronary artery bypass graft.

Exclusion Criteria:

* White blood cell count <3000/mm3
* Platelet count <100,000/mm3
* Hemoglobin <9.0 g/dl
* Creatinine >1.5 mg/dl
* Total bilirubin >1.5 mg/dl
* SGOT, SGPT, or AP >1.5 x upper limit of normal
* Metastatic disease (except peribronchial/hilar lymph nodes=N1 and ipsilateral/subcarinal mediastinal lymph nodes=N2) or malignant pleural effusion detected on preoperative evaluation. Non-malignant effusions are cytology negative, are non-bloody, and are transudates. Effusions visible only on CT and not large enough for safe thoracentesis will not result in ineligibility. Exudative effusions, even if cytologically negative are excluded. Pleural fluid is considered exudative if: the ratio of pleural fluid protein to serum protein is >0.5 or the ratio of pleural fluid LDH to serum to serum LDH >0.6 or Pleural fluid LDH is >200 IU/liter. A staging PET scan will be used to exclude patients. If there are multiple areas of FDG uptake outside the area of the primary tumor and the hilar and ipsilateral mediastinal lymph nodes, the patient will be excluded by virtue of having metastatic disease. If however, only one area shows an increase in FDG uptake, the area of concern will need further evaluation such as a biopsy to exclude metastatic disease.
* N3 lymph nodes (contralateral mediastinal/hilar and supraclavicular/scalene) or T4 primary tumor (malignant pleural effusion or mediastinal invasion) by clinical staging criteria (N3 as seen on CT or PET scan, which may be proven by mediastinoscopy at the investigators discretion).
* Pregnancy.
* Other active malignancy within 2 years with the exceptions of non-melanoma skin cancer and cervical carcinoma in situ.
* Psychologic, familial, sociologic, or geographic conditions, which do not permit biweekly medical follow-up and adherence to the study protocol.
* Prior radiation therapy for any cancer to the thorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Bepler, M.D, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center (now at Karmanos Cancer Institute)
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Journal of Thoracic Oncology: Clinical Efficacy and Predictive Molecular Markers of Neoadjuvant Gemcitabine and Pemetrexed in Resectable Non-small Cell Lung Cancer — http://journals.lww.com/jto/pages/results.aspx?k=bepler%20molecular%20markers&Scope=AllIssues&txtKeywords=bepler%20molecular%20markers

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Surgery Chemotherapy: Pre-Surgery Treatment: Gemcitabine (GemzarR) 1500 mg/m2, and Pemetrexed (AlimtaR) 500 mg/m2. When the chemotherapy treatment was completed, the patient's tumor response was evaluated by a CT scan, pulmonary function test, and another PET scan between days 50 and 63 (during weeks 8 and 9). When there was no growth or spread of the cancer on any of these tests, patients then proceeded to have surgery by week 10 to remove the cancer.
Period: Overall Study
Arm/Group | Pre-Surgery Chemotherapy
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pre-Surgery Chemotherapy
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 31
Age, Continuous [Median (Full Range); unit: years] | 67 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Disease Response - Radiographic
Description: Number of participants with partial or Complete Response. Complete response (CR) is defined as the total disappearance of all malignant and evaluable clinical evidence of cancer without the development of any new malignant lesions documented on the post chemotherapy chest CT and PET scan.
  Partial response (PR) (measurable disease only): When compared with pre-treatment measurements, a reduction of >30% in the sum of the largest diameters of all measurable lesions and absence of new lesions.
Time Frame: 06/20/2008 Index date for patients enrolled between 04/2004 and 04/2006
Population: A radiographic response evaluation was possible in 49 of 52 patients.
Measure: Number; unit: participants
Arm/Group | Pre-Surgery Chemotherapy
Number analyzed (Participants) | 49
participants
  Complete Remission | 1
  Partial Remission | 16

2. Secondary Outcome: Disease Response - Pathologic
Description: Number of participants with Pathologic Complete Response. Pathologic complete response (pCR) is defined by a surgical pathology specimen, which consists of equal to or more than 95% fibrosis and necrosis.
Time Frame: 06/20/2008 Index date for patients enrolled between 04/2004 and 04/2006
Population: A pathologic response evaluation was possible in 43 of 52 patients.
Measure: Number; unit: participants
Arm/Group | Pre-Surgery Chemotherapy
Number analyzed (Participants) | 43
participants | 13 [13 to 43]

3. Secondary Outcome: Survival - Disease Free
Description: Disease-free survival (DFS) is defined as the period of time from surgery to the time when disease recurrence is clearly documented. A histologic confirmation is required in equivalent cases.
Time Frame: 06/20/2008 Index date for patients enrolled between 04/2004 and 04/2006
Population: 40 patients with complete tumor resection.
Measure: Median (Full Range); unit: months
Arm/Group | Pre-Surgery Chemotherapy
Number analyzed (Participants) | 40
months | 33.7 [2.9 to 45.2]

4. Secondary Outcome: Survival - Overall
Description: Median range of number of participants with Overall Survival. Overall survival (OS) will be defined as the period of time from the first day of drug treatment to the date of death of the patient. Patients taken off study will be followed quarterly until death for survival data.
Time Frame: 06/20/2008 Index date for patients enrolled between 04/2004 and 04/2006
Population: All patients
Measure: Median (Full Range); unit: months
Arm/Group | Pre-Surgery Chemotherapy
Number analyzed (Participants) | 52
months | 27.8 [3.8 to 48.6]

5. Secondary Outcome: Toxicity
Description: Number of participants with toxicity ≥ Grade 3 after gemcitabine plus pemetrexed induction chemotherapy.
Time Frame: 06/20/2008 Index date for patients enrolled between 04/2004 and 04/2006
Population: A total of 52 eligible patients, 26 men and 26 women, between the ages of 41 and 83 years received at least one dose of chemotherapy. Only 49 patients were evaluable because 3 patients had only the first cycle.
Measure: Number; unit: participants
Arm/Group | Pre-Surgery Chemotherapy
Number analyzed (Participants) | 49
participants | 18

ADVERSE EVENTS:
Time Frame: 06/20/2008 Index date for patients enrolled between 04/2004 and 04/2006
Description: All Grade 3 and 4 Adverse Events are listed under Serious Adverse Events.
Arm/Group | Pre-Surgery Chemotherapy
Serious Adverse Events (participants affected / at risk) | 18/52
Other Adverse Events (participants affected / at risk) | 1/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Surgery Chemotherapy (N=52)
Alanine Aminotransferase (ALT) - Grade 3 (Metabolism and nutrition disorders) | 3 (3) — > 5.0 <= 20.0
Aspartate Aminotransferase (AST) - Grade 3 (Metabolism and nutrition disorders) | 1 (1) — > 5.0 <= 20.0
Bicarbonate, serum low - Grade 4 (Metabolism and nutrition disorders) | 8 (14) — < 8.0
Dermatology/skin - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1) — Severe
Fatigue - Grade 3 (General disorders) | 1 (1) — Severe fatigue interfering with ADL
Hemoglobin - Grade 3 (Blood and lymphatic system disorders) | 2 (2) — >= 6.5 < 8.
Hyperglycemia - Grade 3 (Metabolism and nutrition disorders) | 7 (21) — > 250.0 <= 500.0
Leukocytes - Grade 3 (Blood and lymphatic system disorders) | 3 (3) — >= 1.0 < 2.
Lymphocytes - Grade 3 (Blood and lymphatic system disorders) | 2 (4) — >= 0.2 < .5
Neutrophils - Grade 3 (Blood and lymphatic system disorders) | 4 (4) — >= 0.5 < 1.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Surgery Chemotherapy (N=52)
Thrombocytopenia - Grade 2 (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No